CLINICAL TRIAL: NCT07044258
Title: Trans-tarsal Stair-step Lateral Extension of the Transconjunctival Approach Versus Transconjunctival Approach in the Management of Orbito-zygomaticomaxillary Complex Fractures (Randomized Controlled Clinical Trial)
Brief Title: Trans-tarsal Stair-step Lateral Extension of the Transconjunctival Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mod-Trans-2/25
Record Dates: First submitted 2025-06-19; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Zygomatic Fractures; Lower Eyelid Entropion
Keywords: Orbito-zygomaticomaxillary Fracture; Transconjunctival Incision; Lower eyelid
MeSH Terms: conditions — Zygomatic Fractures

STUDY DESIGN:
Intervention Model Description: patients presented with oribto-zygomaticomaxillary complex fractures that requires open reduction and internal fixation via trans-tarsal stair-step lateral extension of the transconjunctival approach
Who Masked: Participant
Masking Description: Sequentially numbered, opaque, sealed envelopes (SNOSE) allocation concealment method will be utilized. Each participant included in the study will be given a serial number that will be used in the allocation. These numbers will be written in identical sheets of paper with the group to which each participant is allocated and placed inside opaque envelopes carrying the respective names of participants. A trial independent personnel will be assigned the role of keeping the envelopes and unfolding them only at the time of the operation, so that the participant is allocated to a group which is concealed from the operator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trans-tarsal stair-step lateral extension of the transconjunctival approach (Active Comparator): patients presented with oribto-zygomaticomaxillary complex fractures that requires open reduction and internal fixation via trans-tarsal stair-step lateral extension of the transconjunctival approach
  Interventions: Procedure: trans-tarsal stair-step lateral extension of the transconjunctival approach
- transconjunctival approach (Experimental): patients presented with oribto-zygomaticomaxillary complex fractures that requires open reduction and internal fixation via transconjunctival approach
  Interventions: Procedure: transconjunctival approach

INTERVENTIONS:
Procedure: trans-tarsal stair-step lateral extension of the transconjunctival approach — patients presented with oribto-zygomaticomaxillary complex fractures that requires open reduction and internal fixation via trans-tarsal stair-step lateral extension of the transconjunctival approach
  Arms: trans-tarsal stair-step lateral extension of the transconjunctival approach
Procedure: transconjunctival approach — patients presented with oribto-zygomaticomaxillary complex fractures that requires open reduction and internal fixation via trans-tarsal stair-step lateral extension of the transconjunctival approach
  Arms: transconjunctival approach

SUMMARY:
Open reduction and internal fixation of orbito-zygomaticomaxillary complex (OMC) fractures has challenging impact on the selection of suitable surgical approach to orbital and zygomatic skeleton. Precise repair of the OMC fractures needs a quite understanding of the regional anatomy, precise diagnosis, an accessible exposure and an accurate rigid fixation of fracture to restore the normal form. The esthetic results are one of the most important requirements for this incision in the facial fracture reduction. conventional approaches to the infraorbital rim/orbital floor include (subciliary mid lower eyelid, or subtarsal) and infraorbital incisions. A thorough understanding of each incisional technique requires an appreciation of the relevant anatomy putting in considerations the risk of associated complications. Transconjuctival incision has a lot of advantages, among which is the production of non-visible scar with low incidence of post -operative ectropion and limited access. Trans-tarsal stair-step lateral extension of the transconjunctival approach provides excellent surgical exposure of OMC fractures avoiding the use of a second incision in the area of zygomatic frontal suture. This technique provides good exposure and excellent esthetics.

the aim of this study is to compare Trans-tarsal Stair-Step Lateral Extension of the Transconjunctival approach with transconjunctival approach in the management of orbital and zygomaticomaxillary complex fractures.

DETAILED DESCRIPTION:
This study will be made on twenty patients who will undergo fracture repair of the zygomaticomaxillary complex. Post- operative patient evaluation will be performed with specific attention paid towards accessibility, the exposure duration (time from incision till exposure of the field), esthetic appearance, post- operative pain, postoperative edema, orbital movement, wound healing, scarring, infra orbital nerve sensation and the post- operative ocular complications such as ectropion, entropion, enophthalmos, scleral show and corneal abrasion. Post- operative clinical examinations along with radiographic examination will be done to evaluate the position of zygoma and determine the adequacy of fracture reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with OMC fractures that require open reduction with internal fixation.
2. Patients with orbital wall defects.
3. Patients with blow out fractures.
4. Adult patient between 18 and 60 years with no gender predilections.

Exclusion Criteria:

1. Existing lacerations in the inferior and lateral periorbital regions.
2. Comminuted fracture with bone loss.
3. Existence of infection at the fracture line.
4. Presence of acute or chronic conjunctival diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
exposure duration | During the surgery
  The time taken between performing the incision till exposure of the field will be recorded using a stopwatch.

SECONDARY OUTCOMES:
postoperative edema | 1.5 month
  The postoperative edema will be categorized subjectively into mild (just noticeable), mild to moderate (more obvious edema without occlusion of palpebral fissure), moderate to severe (edema partially occluding palpebral fissure), and severe (edema totally occluding palpebral fissure).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study
Supporting Information: SAP
Access Criteria: to any one who required them after deidentification